CLINICAL TRIAL: NCT00352417
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study of the Effects of VIA-2291, a 5-Lipoxygenase Inhibitor, on Atherosclerotic Plaque and Biomarkers of Vascular Inflammation in Patients With Carotid Stenosis Undergoing Elective Carotid Endarterectomy
Brief Title: Study Effect of VIA-2291 on Atherosclerotic Vascular Inflammation in Patients Undergoing Elective Carotid Endarterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tallikut Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIA-2291-02; 2006-001635-21 (EudraCT Number)
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — atreleuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VIA-2291 (Experimental)
  Interventions: Drug: VIA-2291
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIA-2291 — 100 mg, oral dosing, 1 time daily for 12 weeks
  Other Names: atreleuton
  Arms: VIA-2291
Drug: Placebo — oral dosing, 1 time daily for 12 weeks
  Arms: Placebo

SUMMARY:
This is a study to compare the effect of VIA-2291 vs. Placebo on various inflammatory biomarkers in patients with carotid stenosis scheduled for elective carotid endarterectomy

ELIGIBILITY:
Inclusion Criteria:

* Female patients must be of non-childbearing potential
* Carotid stenosis between 60% and 90% and to be scheduled for CEA surgery
* One or more of the following clinical features: Prior history >4 weeks of cerebrovascular accident (CVA) or transient ischemic attack (TIA) consistent with North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria or prior history of amaurosis fugax occurring at any time
* Diabetes haemoglobin (Hb) A1c between 7.0 and 11% or a history of two or more fasting blood glucose levels >6.9 mmol/L
* Baseline hsCRP >2 mg/L
* Echolucent plaque

Exclusion Criteria:

* Acute CVA or TIA within 4 weeks of enrollment or the presence of ulcerated or unstable plaque requiring urgent carotid endarterectomy
* Renal insufficiency defined as creatinine >1.5 x upper limit of normal (ULN)
* Cirrhosis, recent hepatitis, alanine aminotransferase (ALT) >1 x ULN (i.e., above the normal range) or positive screening test for hepatitis B (hepatitis B surface antigen) or hepatitis C (by ELISA)
* Uncontrolled diabetes mellitus within 1 month prior to study screening, defined as HbA1c >11% at screening
* Congestive heart failure (CHF) defined by the New York Heart Association as functional Class III or IV
* Recent acute coronary syndrome event or coronary artery bypass graft (CABG) surgery (within 4 weeks of enrollment)
* Current atrial fibrillation
* Planned cardiac intervention
* Acetaminophen use in any form in the 7 days before enrollment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — VIA Pharmaceuticals
Locations (3):
- Italy (3):
  - Azienda Ospedali Riuniti Ancona, Ancona
  - Presidio Ospedaliero SS Filippo e Nicola, Avezzano
  - Centro Studi Sull'Invecchiamento, Chieti Scalo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from three Italian Medical Centers
Groups:
- VIA-2291: 100-mg dose
- Matching Placebo: Placebo Dose
Period: Overall Study
Arm/Group | VIA-2291 | Matching Placebo
Started | 24 | 26
Completed | 19 | 21
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Schedule Change | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIA-2291 | Matching Placebo | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 13 | 18 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.86) | 69.5 (8.73) | 68.2 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  Italy | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Cross-sectional Area of Macrophages in Plaque Tissue
Description: Effect of VIA-2291 100-mg relative to placebo after 12 weeks of daily dosing on the percent cross-sectional area of macrophages in plaque tissue using an anti-CD68 antibody
Time Frame: 12 weeks
Population: Evaluable Population with histological sections available
Measure: Mean (95% Confidence Interval); unit: Percent Area
Arm/Group | VIA-2291 | Matching Placebo
Number analyzed (Participants) | 12 | 13
Percent Area | 8.08 [4.3 to 11.9] | 8.19 [3.8 to 12.6]
Statistical Analysis 1: Comparison: VIA-2291 vs Matching Placebo; Test type: Superiority or Other; p = 0.97, t-test, 2 sided; Satterthwaite's method

2. Secondary Outcome: Percent Cross-sectional Area of Anti-5-Lipoxygenase Staining in Plaque Tissue
Description: Effect of VIA-2291 100-mg relative to placebo after 12 weeks of daily dosing on the percent cross-sectional area of anti-5-Lipoxygenase staining in plaque tissue
Time Frame: 12 weeks
Population: Evaluable Population with histological sections available
Measure: Mean (95% Confidence Interval); unit: Percent Area
Arm/Group | VIA-2291 | Matching Placebo
Number analyzed (Participants) | 12 | 13
Percent Area | 1.80 [-0.3 to 3.9] | 0.87 [0.1 to 1.6]
Statistical Analysis 1: Comparison: VIA-2291 vs Matching Placebo; Test type: Superiority or Other; p = 0.37, t-test, 2 sided; Satterthwaite's method

3. Secondary Outcome: Change From Baseline in Whole Blood Leukotriene B4 Production
Time Frame: Baseline and 12 weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | VIA-2291 | Matching Placebo
Number analyzed (Participants) | 16 | 19
pg/ml | -123,000 [-144,000 to -102,000] | -42,900 [-61,900 to -23,900]
Statistical Analysis 1: Comparison: VIA-2291 vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: Change From Baseline in Urine Leukotriene E4 Adjusted for Creatinine
Time Frame: Baseline and 12 Weeks
Population: Evaluable Population
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | VIA-2291 | Matching Placebo
Number analyzed (Participants) | 14 | 14
Percent Change | -64.7 [-75.7 to -48.7] | -15.5 [-41.8 to 22.8]
Statistical Analysis 1: Comparison: VIA-2291 vs Matching Placebo; Test type: Superiority or Other; p < 0.01, ANCOVA; ANCOVA was performed on the natural log transformed data

5. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP)
Time Frame: Baseline and 12 weeks
Population: Evaluable population with both baseline and visit 8 results
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | VIA-2291 | Matching Placebo
Number analyzed (Participants) | 15 | 15
mg/L | -2.0 [-3.1 to -0.9] | 0.2 [-0.9 to 1.3]
Statistical Analysis 1: Comparison: VIA-2291 vs Matching Placebo; Test type: Superiority or Other; p < 0.01, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | VIA-2291 | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 4/24 | 1/26
Other Adverse Events (participants affected / at risk) | 18/24 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIA-2291 (N=24) | Matching Placebo (N=26)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1) | 0 (0)
BENIGN RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VIA-2291 (N=24) | Matching Placebo (N=26)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BLOOD AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD BILIRUBIN UNCONJUGATED INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 3 (3) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 2 (2) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 0/0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GLYCOSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0)
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 0 (0)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The small number, less than optimal quality, and diversity of types of plaque samples posed a significant limitation to the interpretation of the plaque data in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 30 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable.